CLINICAL TRIAL: NCT05929937
Title: No Opioids vs. Minimal Opioids Following Inguinal Hernia Repair
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Clayton Petro (Other)
Responsible Party: Sponsor-Investigator, Clayton Petro, Assistant Professor of Surgery Lerner College of Medicine, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-189
Record Dates: First submitted 2023-06-21; First posted 2023-07-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Pain; Inguinal Hernia
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal | interventions — Analgesics, Opioid

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to receive 5 tablets of Oxycodone (5mg) or none
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Minimal Opioids (Other): Standard of care 5 tablets of Oxycodone (5mg) every 6 hours as needed for pain
  Interventions: Drug: Opioids
- No opioids (Other): Standard of care
  Interventions: Other: No opioids

INTERVENTIONS:
Drug: Opioids — Patients will receive a prescription of 5 tablets of opioids (preferred: Oxycodone, or surgeon preference for Oxycodone intolerance)
  Other Names: Opioid
  Arms: Minimal Opioids
Other: No opioids — Standard of care, patients will not receive a prescription for opioids.
  Arms: No opioids

SUMMARY:
The investigators hypothesize that not prescribing opioids after uncomplicated, outpatient IHR will be non-inferior to prescribing opioids (5 tablets of Oxycodone, 5mg; or surgeon preference for intolerance) with respect to requests for opioid refills. Additionally, the investigators believe there will be no significant difference in postoperative readmission for pain quality of life at 30 days in either group.

DETAILED DESCRIPTION:
Patients presenting with primary or recurrent inguinal hernias, previously repaired in an open fashion, will be considered eligible to be enrolled in this study. Exclusion criteria include patients who cannot tolerate general anesthesia, opioids or NSAIDS, surgeries requiring extensive dissection/hernia sac reduction, or additional procedures, patients requiring inpatient admission postoperatively, and patients who are not able to understand and sign a written consent form. Surgeons will notify a study coordinator at the end of surgery for randomization. Patients will be randomized to opioids versus no opioids at the end of surgery and stratified based on unilateral versus bilateral inguinal hernia repair. The intervention will be not prescribing opioids post-operatively. If patients require prescription for opioids after randomization for uncontrolled pain for the no opioid group, the patient will remain in the intervention group and will be treat as intention to treat which will be recorded in REDCap®. All patients in the study will receive prescriptions for Acetaminophen and Ibuprofen. No other intraoperative or postoperative differences will occur between the two groups.

Baseline information, operative details, and 30-day outcomes are already captured within the ACHQC database, allowing for follow-up, and data capture with decreased effort outside of routine care. Randomization data will be captured and stored in REDCap®.

Baseline patient demographics will be obtained at initial patient recruitment, and baseline ACHQC questionnaires will be completed following patient recruitment. All operative details are already routinely collected and stored in the ACHQC database. Patient-reported quality of life will also be assessed at baseline and at 30 days using the EuraHS Quality Of Life survey tool, which is collected for all patients entered into the ACHQC as part of the ACHQC Inguinal Hernia Postoperative Assessment. Patients will be required to complete these forms at each clinic visit, or via telephone contact, as this is standard procedure for all patients entered into the ACHQC. At the time of the one-month follow-up clinic visits, a routine physical examination will be performed on all patients.

Outcomes to be investigated:

* Specific Aim #1: To determine if the use of post-operative use of opioids results in a difference in rate of opioid refills/requests when compared to those not initially prescribed opioids.
* Specific Aim #2: To determine if the use of post-operative use of opioids results in a difference in Patient-Reported Outcome Measurement Information System (PROMIS Pain Intensity) scores at the 1 month follow up visit post-operatively when compared to those not prescribed opioids.
* Specific Aim #3: To determine if the use of post-operative use of opioids results in a difference in EuraHS (European registry for abdominal wall hernias) Quality of Life (QoL) scores at the 1 month follow up visit post-operatively when compared to those not prescribed opioids.
* Specific Aim #4: To determine if the use of post-operative use of opioids results in a difference in all 30-day complications when compared to those not prescribed opioids.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 years or older
* Patients undergoing elective unilateral or bilateral inguinal hernia repairs
* Patients able to tolerate general anesthesia

Exclusion Criteria:

* Patients who cannot tolerate general anesthesia,
* Patients who cannot tolerate opioids or NSAIDS,
* Patients on opioids for chronic pain management (defined as near daily use within 90 days),
* Patients who undergo surgeries requiring extensive dissection/hernia sac reduction, or additional procedures,
* Patients requiring inpatient admission postoperatively
* Patients who are not able to understand and sign a written consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 904 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Opioid refills/requests | At the one month follow up visit
  The number of opioid prescription refills/requests will be compared between the two groups

SECONDARY OUTCOMES:
Postoperative pain | At the one month follow up visit
  Postop pain will be assessed using the Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity 3a scale scale between the two groups where higher scores mean worse pain
Quality of life, pain, cosmesis | At the one month follow up visit
  Quality of life, pain, and cosmetic outcomes will be assessed using the EuraHS (European registry for abdominal wall hernias) Quality of Life scale between the two groups where higher scores mean worse quality of life.
Patient satisfaction | At the one month follow up visit
  Overall patient satisfaction: patients will be asked if they are dissatisfied, neutral, or satisfied with respect to their postoperative pain management and the responses will be compared between the two groups
Number of emergency room (ER)/clinic/urgent care visits for pain | At the one month follow up visit
  The number of emergency room/clinic/urgent care visits for pain will be compared between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Clayton C Petro, MD, Principal Investigator — The Cleveland Clinic
Locations (8):
- United States (7):
  - MemorialCare, Fountain Valley, California
  - Corewell Health, Royal Oak, Michigan
  - University Hospitals, Cleveland, Ohio
  - Cleveland Clinic Center for Abdominal Core Health, Cleveland, Ohio
  - Prisma Health, Greenville, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- North York General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No